CLINICAL TRIAL: NCT07012005
Title: A Phase 1, Open-label, Parallel-group Study to Assess the Pharmacokinetics, Safety, and Tolerability of BPN14770 in Participants With Severe Renal Impairment and Healthy Control Participants
Brief Title: Study of BPN14770 in Participants With Severe Renal Impairment and Healthy Controls
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2415A4113
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — BPN14770

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Participants With Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single dose of BPN14770 administered orally in the fasted state on Day 1.
  Interventions: Drug: BPN14770
- Group 2: Participants With Normal Renal Function (Experimental): Participants with normal renal function will receive a single dose of BPN14770 administered orally in the fasted state on Day 1.
  Interventions: Drug: BPN14770

INTERVENTIONS:
Drug: BPN14770 — BPN14770 will be administered per schedule specified in the arm description.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), safety, and tolerability of BPN14770 in participants with severe renal impairment and those with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Considered to be healthy (for healthy participants) or medically stable (for participants with renal impairment), as determined by medical evaluation including medical/surgical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiogram (ECG) during the screening period and upon admission to the clinical research unit (CRU).
* Body weight ≥ 50 kilograms (kg) and body mass index (BMI) within the range 18.5 to <40.0 kg/square meter (m^2) (inclusive)

Participants With Renal Impairment:

* Participants that are not undergoing hemodialysis and have severe renal impairment based upon their 2021 chronic kidney disease epidemiology collaboration (CKD-EPI) creatinine formula creatinine clearance estimate (CLcr) estimated glomerular filtration rate (eGFR) estimate and the participant's body surface area (BSA) calculated at the screening visit

  a. Severe renal impairment: eGFR <30 milliliters (mL)/minute (min)
* A stable medication regimen is required, defined as not starting new drug(s) or changing dosage(s) within 14 days prior to administration of study intervention through the follow-up/early termination visit.

Healthy Participants:

* Participants with clinical laboratory tests within normal reference range for the laboratory, or abnormal but considered not clinically significant by the investigator. Renal function, calculated by 2021 CKD-EPI creatinine formula and the participant's BSA, must be normal (that is, eGFR ≥90 mL/min)
* Matched to each participant with severe renal impairment with respect to sex, age (± 10 years), and BMI (± 10%)

Exclusion Criteria:

All Participants:

* History or presence of/significant history of or current cardiovascular, respiratory, renal, gastrointestinal (GI), endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data in the judgement of the investigator
* Current or chronic history of liver disease or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones)
* History of GI surgery including but not limited to gastric resection and/or intestinal resection that resulted in a clinically significant abnormality in GI function
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Participants with fluctuating or rapidly deteriorating renal function. Assessment of the stability of the participant's renal function will be determined by the investigator.
* Any condition requiring medication and/or other treatment other than protocol-specified medication for participants with renal impairment, such as dietary restriction and physical therapy
* Participant with poor venous access
* History of Coronavirus Disease 2019 (COVID-19) infection within 14 days prior to the screening visit or admission to the CRU, or close contact with a COVID-19 patient in the 14 days prior to the screening visit or admission to the CRU as reported by the participant and the participant's medical history.
* Sensitivity to the study intervention, or components thereof, or a drug or other allergy, including food allergy, that in the opinion of the investigator or medical monitor contraindicates participation in the study.

Participants With Renal Impairment:

* Participant with acute renal failure or a kidney transplant history or requiring renal dialysis during the study period
* Current or anticipated need for hemodialysis during the study

NOTE: Other protocol-specified inclusion and exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of BPN14770 | 0 (predose) up to 240 hours postdose on Day 1 to Day 11
Time to Reach Cmax (Tmax) of BPN14770 | 0 (predose) up to 240 hours postdose on Day 1 to Day 11
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration After Dosing (AUC0-last) of BPN14770 | 0 (predose) up to 240 hours postdose on Day 1 to Day 11

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 15

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida